CLINICAL TRIAL: NCT04376723
Title: Mental Health Mobile Application Self-Help for Adolescents Exhibiting Mild Psychological Distress: A Single Case Experimental Design
Brief Title: Mental Health Apps for Mild Psychological Distress Amongst Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: Lincolnshire Partnership NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20010
Record Dates: First submitted 2020-03-19; First posted 2020-05-06 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-04

CONDITIONS: Psychological Distress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assisted self-guidance (Experimental): Participants will be asked to use the app for five weeks and will be contacted via telephone once a week by a researcher to provide a rationale for using the app, or to offer any information about the app itself. This will not be used to provide therapeutic intervention.
  Interventions: Other: Mental Health Mobile Application

INTERVENTIONS:
Other: Mental Health Mobile Application — Mobile phones will not be provided to participants, but app subscriptions will be provided.

SUMMARY:
This study investigates mental health mobile apps, to understand their efficacy in reducing mild levels of psychological distress amongst adolescents. All participants will be provided with an app which is already available in the public domain, and will be asked to use the app for guided self-help. Half of participants will receive a weekly telephone call, whilst the other half will not.

DETAILED DESCRIPTION:
The subscription version of the app "Sanvello" has several self-help exercises based on Cognitive Behavioural Therapy (to identify and challenge their thinking styles) and Mindfulness practices (to connect them with the present moment). Participants will be asked to complete these exercises on a daily basis for five weeks.

Telephone calls will be provided weekly to half of participants to provide information about the app, or a rationale for its use. This phone call will not serve to provide any extra intervention or therapy to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 13-18 years, as the proposed research aims to investigate "adolescents".
* Have capacity to give informed consent, to ensure the integrity of participants and prioritise their best interests.
* Be awaiting input from the Healthy Minds Lincolnshire service, given the method of recruitment, prospective participants will be on a waiting list for the named service.
* Be experiencing psychological distress, to fulfil the research aims.

Exclusion Criteria:

* Accessing crisis support, to ensure that necessary support is not being withheld due to research participation.
* They do not speak and understand English, to ensure the app-intervention and measures (which are in English) may be completed, and so interviews may be conducted without a translator.
* They are unable to access or use a smart device, the internet, and the app, as they must be able to access a device daily and be technology literate to utilise the intervention.
* For 13-15 year olds: parental consent must also be provided to take part. If this is not provided, they will be unable to participate. Those aged 16-18 years can provide consent for themselves.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Kessler 10 | Through study completion, an average of 18 weeks
  10 item self-report measure of psychological distress with five response categories (none of the time, a little of the time, some of the time, most of the time, all of the time). Scores range from 10 to 50; a higher score indicates more psychological distress.
Cognitive Emotion Regulation Questionnaire-Short | Through study completion, an average of 18 weeks
  18 item self-report process measure of cognitive strategies to regulate emotions with five response categories (almost never, rarely, occasionally, frequently, almost always). This measure has nine subscales, with two items each (self-blame, acceptance, rumination, positive refocusing, refocus on planning, positive reappraisal, putting into perspective, catastrophising, other-blame). Scores per subscale range from 2 to 10; higher scores indicate greater use of specific cognitive strategies, some of which are favourable and others indicate negative thinking styles.

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale | Through study completion, an average of 18 weeks
  14 item self-report measure of wellbeing with five response categories (none of the time, rarely, some of the time, often, all of the time). Scores range from 14 to 70; a higher score indicates better mental wellbeing and scores below a cut point of 40 indicate low wellbeing.
CompACT-8 | Through study completion, an average of 18 weeks
  8 item self-report measure of psychological flexibility with six response categories (strongly disagree, moderately disagree, slightly disagree, neither agree nor disagree, slightly agree, moderately agree, strongly agree). Total scores range from 0 to 48, with higher scores indicating greater psychological flexibility. This measure has three subscales: openness to experience (range of scores: 0 to 18), behavioural awareness (range of scores: 0 to 12), and valued action (range of scores: 0 to 18); as with the overall score, higher subscale scores indicate favourable outcomes.

OTHER OUTCOMES:
Personal Questionnaire | Through study completion, an average of 18 weeks
  Participant-generated goals, established by asking each participant which difficulties the individual would like to work on. Ten items are established with each participant (e.g. with a focus on symptoms, mood, specific activities, relationships, or self-esteem). Each of the ten items is rated according to seven response categories (this has bothered me: not at all, very little, little, moderately, considerably, very considerably, maximum possible). Scores range between 10 and 70, with higher scores indicating greater difficulties.
Change Interview | Up to 18 weeks
  Participant view of change according to a semi-structured interview of ten key questions.

CONTACTS AND LOCATIONS:
Overall Officials: David Dawson, DClinPsy, Study Chair — University of Lincoln
Locations (1):
- Lincolshire Partnership NHS Foundation Trust, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grist R, Porter J, Stallard P. Mental Health Mobile Apps for Preadolescents and Adolescents: A Systematic Review. J Med Internet Res. 2017 May 25;19(5):e176. doi: 10.2196/jmir.7332. PMID 28546138
- [Derived] Badesha K, Wilde S, Dawson DL. Mental health mobile application self-help for adolescents exhibiting psychological distress: A single case experimental design. Psychol Psychother. 2023 Mar;96(1):223-248. doi: 10.1111/papt.12436. Epub 2022 Nov 7. PMID 36345016